CLINICAL TRIAL: NCT01645176
Title: Hydroxychloroquine/Atorvastatin in the Treatment of OA of the Knee
Brief Title: Hydroxychloroquine/Atorvastatin in the Treatment of Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Mark Genovese, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23784
Record Dates: First submitted 2012-05-31; First posted 2012-07-20 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis of the Knee
Keywords: OA; Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hydroxychloroquine; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxychloroquine/Atorvastatin open label (Experimental)
  Interventions: Drug: Hydroxychloroquine/Atorvastatin

INTERVENTIONS:
Drug: Hydroxychloroquine/Atorvastatin — Hydroxychloroquine 200-600 mg /day Atorvastatin 40 mg/day

SUMMARY:
The purpose of this study of a combination therapy of hydroxychloroquine and atorvastatin is to learn about the effects in inflammation and pain in patients with Osteoarthritis of the knee. These medications are FDA approved and commercially available.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory subjects with OA of the knee with symptoms for at least 6 months and pain on the majority of days in the last 30 days. Symptoms must include knee joint pain.
2. Male or female adults age >40 years with a body mass index <35
3. Radiographic evidence of at least one osteophyte in either knee on posteroanterior (PA) and lateral standing, flexed x-ray.
4. A Kellegren-Lawrence score of 2-3, or KL score of 1 accompanied by a clinically apparent effusion in the index knee.
5. A WOMAC pain score of >8 on the index knee at screening visit.

Exclusion Criteria:

1. A requirement for treatment with high potency opioids for pain relief.
2. Unwilling to abstain from NSAIDs and/or other analgesic medications except acetaminophen (i.e., COX-2 inhibitors, tramadol) for 48 hours and acetaminophen for 24 hours prior to pain assessments during the study. Subjects taking low dose aspirin for cardiovascular health may remain on their stable dose throughout the study.
3. On an unstable dose of NSAIDs or analgesics for at least 1 months prior to screening visit 1.
4. Using a handicap assistance device (i.e., cane, walker) >50% of the time.
5. Undergoing new physical therapy or participating in a weight loss or exercise program that has not been stable for at least 3 months prior to screening visit 1 and will not remain stable during their participation in the study.
6. Had a previous history of arthroscopic or open surgery to the index knee in the past 6 months or planned surgery during study follow up.
7. Had joint replacement surgery in the index knee.
8. Received corticosteroid, short acting hyaluronic acid, or other intraarticular injections of the index knee within 3 months of screening visit 1 and/or not willing to abstain from treatments for the duration of the study
9. A history in the past 5-10 years of reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis, amyloidosis or fibromyalgia.
10. Clinical signs and symptoms of active knee infection or radiographic evidence of crystal disease other than chondrocalcinosis (i.e. gout).
11. A history of abnormal laboratory results >2.5 x ULN indicative of any significant medical disease, which in the opinion of the investigator, would preclude the subjects participation in the study
12. Any of the following abnormal laboratory results during screening:

    * ALT and/or AST >2.5x ULN
    * Hemoglobin <9 g/dL
    * WBC <3500 cells/mm3
    * Lymphocyte count <1000 cells/mm3
    * Serum creatinine >1.5 x ULN or calculated Glomerular filtration rate less than 50.
    * Creatine phosphokinase level > 2x ULN
13. A history of malignancy in the past ten years (<10 years), with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ.
14. Significant hip pain, ipsilateral to the index knee that may interfere with assessments of index knee pain
15. A known or clinically suspected infection with human immunodeficiency virus (HIV), or hepatitis C or B viruses
16. Participated within 3 months or will participate concurrently in another investigational drug or vaccine study
17. A history of drug or alcohol dependence or abuse in the past 3 years
18. A female with reproductive capability who is unwilling to use birth control for the duration of the study and/or intends to conceive within 12 months of dosing.
19. Ongoing use of hydroxychloroquine, or any anti-malarial, or prior history of use within past 3 months or any prior history of history of allergy, hypersensitivity or toxicity to antimalarial use.
20. Ongoing use of a statin (HMG Co A reductase inhibitor), or use within past 3 months or any prior history of history of allergy, hypersensitivity, or toxicity to statin use.
21. Use of fibric acid derivative in past 3 months.
22. Other serious, non-malignant, significant, acute or chronic medical or psychiatric illness that, in the judgment of the investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Responders to ad in local paper, medical clinic May 2012 - Dec 2014
Pre-assignment Details: Osteoarthritis of knee
Units Other Than Participants: knee
Period: Overall Study
Arm/Group | Hydroxychloroquine/Atorvastatin Open Label
Started | 21; 21 knee
Completed | 16; 16 knee
Not Completed | 5; 5 knee
Not completed — Lack of Efficacy | 4
Not completed — did not complete final MRI | 1

BASELINE CHARACTERISTICS:
Population: Osteoarthritis of knee
Arm/Group | Hydroxychloroquine/Atorvastatin Open Label
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 64.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 16
WOMAC PAIN [Mean (Standard Deviation); unit: units on a scale] — (WOMAC) The Western Ontario and McMaster Universities Osteoarthritis Index
  Rates activities for Stiffness, Pain and Physical Function according to the following:
  scale of difficulty: 0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely
  units on a scale | 9.8 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Synovitis
Description: MRI readings performed independently by two musculoskeletal radiologists, using a semi-quantitative scoring system based on MRI assessment of knee OASynovitis scored using axial & sagittal CE-MRI sequence, while effusion & bone marrow lesions were scored using non-CE-MRI sequences of parent study.
  Synovitis defined as enhancing thickened synovium (>2 mm) & was evaluated at nine sites of joint-medial & lateral parapatellar recess, suprapateller, infrapatellar, intercondylar, medial & lateral perimeniscal, & adjacent to anterior & posterior cruciate ligaments (ACL/PCL) in all subjects. Synovial thickness was scored semi-quantitatively based on maximal thickness in any slice at each site as follows: grade 0 if <2mm, grade 1 if 2-4 mm & grade 2 if >4mm. For assessment of whole knee synovitis scores of all sites were summed and categorized: 0-4 normal or equivocal synovitis; 5-8 mild synovitis; 9-12 moderate synovitis & >/= 13 severe synovitis.
Time Frame: baseline and 16 weeks
Population: Participants with osteoarthritis of knee
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Osteoarthritis of Knee: Change in MRI synovitis
Arm/Group | Osteoarthritis of Knee
Number analyzed (Participants) | 16
units on a scale | 9.8 (4.4)

ADVERSE EVENTS:
Time Frame: monthly for 4 months
Description: All subjects were monitored for AEs during the study. Assessments included monitoring of any or all of the following parameters: the subject's clinical symptoms; laboratory, pathological, radiological, or surgical findings; physical examination findings; or other appropriate tests and procedures.
Arm/Group | Hydroxychloroquine/Atorvastatin Open Label
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No